CLINICAL TRIAL: NCT04104542
Title: MOCHI: A Randomized Controlled Trial of Mindfulness as a Treatment for Chronic Pelvic Pain in Active Duty Women
Brief Title: MOCHI: An RCT of Mindfulness as Treatment for Chronic Pelvic Pain in AD Women
Acronym: AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Carol Crisp, Principal Investigator, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 18-078
Record Dates: First submitted 2019-05-01; First posted 2019-09-26 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pelvic Pain; Depression; Inflammation Pelvic
Keywords: military; chronic pelvic pain; inflammation; mindfulness
MeSH Terms: conditions — Depression; Pelvic Inflammatory Disease; Inflammation | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness MTHM (Experimental): online mindfulness based stress reduction training
  Interventions: Behavioral: Mindfulness based stress reduction
- Mindfulness JBSA (Experimental): online mindfulness based stress reduction training
  Interventions: Behavioral: Mindfulness based stress reduction
- Healthy Lifestyle MTHM (Sham Comparator): online healthy lifestyle training
  Interventions: Behavioral: Healthy Lifestyle
- Healthy Lifestyle JBSA (Sham Comparator): online healthy lifestyle training
  Interventions: Behavioral: Healthy Lifestyle

INTERVENTIONS:
Behavioral: Mindfulness based stress reduction — on-line training on the website = www.palousemindfulness.com
  Other Names: MBSR
  Arms: Mindfulness JBSA; Mindfulness MTHM
Behavioral: Healthy Lifestyle — Diet and Exercise
  Other Names: HL
  Arms: Healthy Lifestyle JBSA; Healthy Lifestyle MTHM

SUMMARY:
Subject Population: Active duty (AD) women with chronic pelvic pain (CPP) have different demands and stressors placed on them compared with their civilian counterparts. Due to a decrease in functionality from pain, not addressing these women's untreated CPP could be detrimental in readiness missions. With limited studies on AD women with CPP or sufficient treatments available, this study seeks to compare the effects on pain, depression, and inflammation in the mindfulness-based stress reduction (MBSR) group with a self-paced Healthy Lifestyle (HL) education control.

Research Design: This randomized controlled trial will compare depression, pain, and biomarkers known for inflammation and pain in AD women with CPP pre-post an 8-week MBSR online intervention (n=55) with a self-directed Healthy Lifestyle control (n=55).

Instruments: All participants will complete a demographic worksheet, Five Facets of Mindfulness Questionnaire (FFQ), a brief pain inventory (BPI), and a Patient Health Questionnaire (PHQ-9) pre-post intervention (MBSR or HL).

Procedure: Participants will have 8-weeks of online training with voice-over slides in RedCap. The primary investigator will contact participants weekly for both groups and review diaries to help monitor fidelity and guide progress. Blood will be drawn for biomarkers for inflammation and pain and questionnaires will be completed pre-post intervention.

DETAILED DESCRIPTION:
The Purpose of this randomized controlled trial (RCT) is to compare the effects of an 8-week on-line MBSR training program with a HL self-directed education program (control) on pain, depression, and inflammation using questionnaires and biomarkers in AD women with CPP.

Specific Aims and Research Questions It is important to understand predictors of CPP among women in active military service and test strategies that may mitigate the negative impact of CPP. The long-term goal of this research is to identify a non-invasive, easy to learn, alternative method that can successfully assist active duty women with CPP to regulate daily perceptions of their body, improve pain management skills to better cope, and ultimately improve functionality and QOL.

Specific Aim #1: To compare the depression of active duty (AD) women with CPP pre-post an 8-week online MBSR program with an 8-week Healthy Lifestyle (HL) nutrition self-paced education.

Hypothesis #1: AD women with CPP in an 8-week MBSR Program will have an overall decreased depression pre-post as compared to the HL control.

Question #1: What is the effect of an online MBSR training program as compared to a HL control pre-post on AD women's depression scores? Specific Aim #2: To compare the perception of pain in AD women with CPP pre-post an 8-week online MBSR program with an 8-week HL control.

Hypothesis 2: AD women with CPP in an 8-week MBSR Program will have overall decreased perception of pain pre-post as compared to the HL control.

Question #2: What is the effect of an online MBSR training program as compared to a HL control pre-post on AD women's perception of pain? Specific Aim #3: Compare the inflammatory biomarkers and miRNAs changes in AD women with CPP pre-post an 8-week online MBSR program with an 8-week HL control.

Hypothesis #3: AD women with CPP in an 8-week MBSR training program will demonstrate an overall decrease in inflammation as demonstrated by the biomarker changes pre-post.

Question #3: What is the effect of an online MBSR training program as compared to a HL control pre-post on active duty women's inflammatory biomarkers?

ELIGIBILITY:
Inclusion Criteria:

* 21-50 years of age
* active duty female
* English as first language
* diagnosed with chronic pelvic pain
* Has access to a computer, telephone, and wifi
* Will not PCS or deploy in the next 3 months without access to computer
* consent form signed

Exclusion Criteria:

* abdominal or pelvic surgery in last 6 months
* known vaginal or pelvic infection at the time of study enrollment, not currently being treated
* menopausal
* pregnant
* breastfeeding
* underlying disease including: diabetes, tumors, auto-immune disorders

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Active Duty Female
Enrollment: 41 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory Questionnaire measuring participants pelvic pain | pre- and at the end of the intervention (6 weeks)
  Brief Pain Inventory - Short Form (BPI-sf) is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on their daily functioning. The participant rates their worst, least, average, and current pain intensity, lists current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10 point scale. The BPI-sf is a modification of the Brief Pain Inventory - Long Form. Pelvic pain as measured by the Brief Pain Inventory questionnaire for each participant before the interventions and at 6 weeks. The BPIsf assesses severity of pain (4 items) and the impact of pain on daily function (7 items). Self-report Likert type scale measuring from no pain (0) to maximum pain (10).

SECONDARY OUTCOMES:
Five Facets of Mindfulness Questionnaire measuring mindfulness | pre- and at the end of the intervention (6 weeks)
  The Five Facets of Mindfulness questionnaire will be used to measure mindfulness for each participant before and at the end of the intervention. This scale has sub-scales that measure observing, describing, acting with awareness, and accepting without judgement which are combined for a total score. Self-report scale using 0=never/rare to 5=very often to always true for each question.
Patient Health Questionnaire -9 (PHQ-9) measuring depression | pre- and at the end of the intervention (6 weeks)
  The PHQ-9 will be used to measure depression before and at the end of the interventions using a self-rated Likert type scale. The 9 item questionnaire asks participants to rate how often they experience depression and somatic complaints over the last 2 weeks. A consistent cut-off score for the PHQ-9 includes scores of 5 (mild), 10 (moderate), 15 (moderately severe), and 20 (severe) depression.
Inflammation changes as measured in ng/ml of Interluekin-8, Interleukin 1ra, and Tumor Necrosis Factor-a pre- and post- intervention (6 weeks)/Physiologic parameter | pre- and at the end of the intervention (6 weeks)
  Elisa's were used to measure changes in inflammation using ng/ml before and after interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Carol D Crisp, PhD (c), Principal Investigator — University of Missouri, Kansas City
Locations (1):
- Univeristy of Missouri-Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crisp CD, Baldi R, Fuller M, Abreu E, Nackley AG. Complementary Approaches for Military Women with Chronic Pelvic Pain: A Randomized Trial. J Integr Complement Med. 2023 Jan;29(1):22-30. doi: 10.1089/jicm.2022.0616. Epub 2022 Oct 12. PMID 36251868